CLINICAL TRIAL: NCT00895934
Title: A Phase 1/2 Study of Vorinostat (Zolinza®) in Combination With Gemtuzumab Ozogamicin (Mylotarg®) and Azacitidine (Vidaza®) in Patients 50 Years of Age and Older With Relapsed/Refractory Non-APL Acute Myeloid Leukemia (AML)
Brief Title: Vorinostat, Azacitidine, and Gemtuzumab Ozogamicin for Older Patients With Relapsed or Refractory AML
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01147; NCI-2012-01147 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IR-6921 (Other: Fred Hutchinson Cancer Research Center); CDR0000642213 (Other: FDA Center for Drug Research); 2288.00 (Other: Fred Hutchinson Cancer Research Center); 8297 (Other: CTEP); P30CA015704 (NIH)
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Results first posted 2015-02-06 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Vorinostat; Gemtuzumab; Calicheamicins; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1 - Dose Finding (Experimental): Varying schedules and dose levels of vorinostat, azacitidine and gemtuzumab ozogamicin. Includes cohorts 1-3.
  Interventions: Drug: vorinostat; Drug: gemtuzumab ozogamicin; Drug: azacitidine
- Phase 2 - Treatment at Selected Dose (Experimental): Vorinostat 400 mg/day on days 1-9, azacitidine 75 mg/m2/day on days 1-7, gemtuzumab ozogamicin 3 mg/m2/day on days 4 and 8.
  Interventions: Drug: vorinostat; Drug: gemtuzumab ozogamicin; Drug: azacitidine

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: gemtuzumab ozogamicin — Given intravenously (IV)
  Other Names: Calicheamicin; CDP-771; CMA-676; Mylotarg
Drug: azacitidine — Given IV or subcutaneously (SC)
  Other Names: 5-AC; 5-azacytidine; azacytidine; Vidaza

SUMMARY:
The purpose of this study is to test the safety of vorinostat (Zolinza) and azacitidine (Vidaza) when combined with gemtuzumab ozogamicin (GO) at different dose levels. These drugs increase the effect of GO against leukemia cells in the test tube, but we don't know yet whether they also increase the anti-leukemia effect of GO in people.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the vorinostat dose with the most favorable efficacy and toxicity when combined with azacitidine and GO.

SECONDARY OBJECTIVES:

I. Describe the complete response (CR)/ CR with inadequate recovery (CRi) rate after a total of 6 cycles of therapy.

II. Describe the disease-free survival of patients that achieve CR/CRi. III. Determine whether acute myeloid leukemia (AML) characteristics associated with preclinical GO efficacy predict for clinical benefit, and assess whether differentiation-inducing agents modulate these characteristics and lower the apoptotic threshold for calicheamicin-gamma1-induced cytotoxicity (in vitro correlative and mechanistic studies).

OUTLINE: This is phase I, dose-escalation study of vorinostat followed by a phase II study.

Patients receive vorinostat orally (PO) on days 1-9, azacitidine subcutaneously (SC) or intravenously (IV) over 10-40 minutes on days 1-7, and gemtuzumab ozogamicin IV over 2 hours on day 4 and 8. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Prior morphological diagnosis of acute myeloid leukemia (AML) other then acute promyelocytic leukemia (APL) according to the 2001 WHO criteria; patients with biphenotypic AML are eligible
* Need for first salvage chemotherapy for persistent or relapsing disease, defined by standard criteria, after at least one course of conventional chemotherapy
* A bone marrow biopsy is not required but should be obtained if the aspirate is dilute, hypocellular, or not aspirable; outside marrow exams performed within the stipulated time period are acceptable if the slides are reviewed at the study institution
* Flow cytometric analysis of the marrow aspirate per institutional practice guidelines
* Duration of first complete remission (CR1) < 12 months (or primary resistant disease)
* Patients with prior autologous or allogeneic hematopoietic cell transplantation (HCT) if relapse occurs 6-12 months post-transplant
* ECOG/WHO/Zubrod performance status of 0-3 within 14 days prior to registration
* Off any active therapy for AML except hydroxyurea for at least 14 days prior to study registration, with resolution of all grade 3 and 4 non-hematological toxicities
* Willingness to discontinue taking any medications known to cause a risk of Torsades de Pointes
* Bilirubin =< 1.5 x Institutional Upper Limit of Normal (IULN) unless elevation is due to hepatic infiltration by AML, Gilbert's syndrome, or hemolysis (within 7 days prior to registration)
* SGOT (AST) and SGPT (ALT) =< 1.5 x IULN unless elevation is due to hepatic infiltration by AML (within 7 days prior to registration)
* Serum creatinine =< 1.5 x IULN (within 7 days prior to registration)
* No clinical or radiographical evidence of heart failure
* white blood cell (WBC) < 25,000/uL within 3 days prior to registration
* Patients with symptoms/signs of hyperleukocytosis or WBC > 100,000/uL can be treated with leukapheresis prior to enrollment
* Collection of bone marrow and peripheral blood specimens for correlative studies prior to study treatment is highly recommended; peripheral blood only is acceptable if the peripheral blast count is > 5,000/uL and > 50% of total WBC
* Must agree to use adequate contraception prior to and during the study
* Can understand and sign a written informed consent document; a legally authorized representative can provide consent if the patient is unable

Exclusion Criteria:

* Remission or second or later relapse
* Diagnosis of another malignancy, unless diagnosed at least 2 years earlier and disease-free for at least 6 months after completion of curative intent therapy except:

  * Treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, if definitive treatment has been completed
  * Organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values if hormonal therapy has been initiated or a radical prostatectomy was performed
* Refractory/relapsing blast crisis of chronic myeloid leukemia (CML)
* Prior anti-AML treatment with GO, histone deacetylase (HDAC) inhibitor (including the use of valproic acid for control of seizure activity or other purposes), or demethylating agent
* Known hypersensitivity to GO, vorinostat, azacitidine, or mannitol
* Possible central nervous system (CNS) involvement with leukemia unless a lumbar puncture confirms no leukemic blasts in the cerebralspinal fluid (CSF)
* HIV-positive patients with cluster of differentiation (CD)4 count is < 200 cells/uL or if AIDS-related complications
* Pregnancy; breastfeeding should be discontinued if the mother is treated with vorinostat, azacitidine, and GO
* Uncontrolled systemic infection, despite appropriate antibiotics or other treatment)
* Receipt of any other investigational agents

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-05; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Walter, Principal Investigator — Fred Hutchinson Cancer Center
Locations (4):
- United States (4):
  - Stanford University Hospitals and Clinics, Stanford, California
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Walter RB, Medeiros BC, Gardner KM, Orlowski KF, Gallegos L, Scott BL, Hendrie PC, Estey EH. Gemtuzumab ozogamicin in combination with vorinostat and azacitidine in older patients with relapsed or refractory acute myeloid leukemia: a phase I/II study. Haematologica. 2014 Jan;99(1):54-9. doi: 10.3324/haematol.2013.096545. Epub 2013 Oct 18. PMID 24142996

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Azacitidine 75mg/m^2/day, days 1-7, Vorinostat 200mg/day, days 1-9; and Gemtuzumab Ozogamicin 3mg/m^2, Day 8 only. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Vorinostat: Given orally
  Gemtuzumab ozogamicin: Given IV
  Azacitidine: Given IV or SC
  laboratory biomarker analysis: Correlative studies
- Dose Level 2: Patients receive Azacitidine 75mg/m^2/day, days 1-7, Vorinostat 300mg/day, days 1-9; and Gemtuzumab Ozogamicin 3mg/m^2, Day 8 only. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Vorinostat: Given orally
  Gemtuzumab ozogamicin: Given IV
  Azacitidine: Given IV or SC
  laboratory biomarker analysis: Correlative studies
- Dose Level 3: Patients receive Azacitidine 75mg/m^2/day, days 1-7, Vorinostat 400mg/day, days 1-9; and Gemtuzumab Ozogamicin 3mg/m^2, Day 8 only. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Vorinostat: Given orally
  Gemtuzumab ozogamicin: Given IV
  Azacitidine: Given IV or SC
  laboratory biomarker analysis: Correlative studies
- Dose Level 4: Patients receive Azacitidine 75mg/m^2/day, days 1-7, Vorinostat 400 mg/day, days 1-9; and Gemtuzumab Ozogamicin 3mg/m^2, Days 4 and 8. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Vorinostat: Given orally
  Gemtuzumab ozogamicin: Given IV
  Azacitidine: Given IV or SC
  laboratory biomarker analysis: Correlative studies
Period: Dose Escalation
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Started | 3 | 3 | 3 | 6
Completed | 3 | 3 | 3 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Efficacy of Most Tolerated Dose
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Started | 0 | 0 | 0 | 37
Completed | 0 | 0 | 0 | 37
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 Dose-Finding Cohorts 1-3: Patients receive vorinostat PO on days 1-9, azacitidine SC or IV over 10-40 minutes on days 1-7, and gemtuzumab ozogamicin IV over 2 hours on day 8. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  vorinostat: Given orally
  gemtuzumab ozogamicin: Given IV
  azacitidine: Given IV or SC
  laboratory biomarker analysis: Correlative studies
- Phase 2/Selected Dose: Azacitidine 75 mg/m2 SC or IV on days 1-7, vorinostat 400 mg qd po on days 1-9, gemtuzumab ozogamicin 3 mg/m2 IV on days 4 and 8. Includes cohort 4 from the Phase 1 portion of the study. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose-Finding Cohorts 1-3 | Phase 2/Selected Dose | Total
Number analyzed (Participants) | 9 | 43 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 21 | 25
  >=65 years | 5 | 22 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 18 | 23
  Male | 4 | 25 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 6 | 40 | 46
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 6 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 34 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 43 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicity (Phase I)
Time Frame: 42 days
Measure: Number; unit: participants
Groups:
- Dose 1: Vorinostat 200, D8
- Dose 2: Vorinostat 300, D8
- Dose 3: Vorinostat 400, D8
- Dose 4: Vorinostat 400, D4 and D8
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4
Number analyzed (Participants) | 3 | 3 | 3 | 6
participants | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Dose-limiting Toxicity After the Vorinostat Dose
Time Frame: Up to 3 years
Measure: Number; unit: participants
Groups:
- Phase 2/Selected Dose: Azacitidine 75 mg/m2 on days 1-7, vorinostat 400 mg qd on days 1-9, gemtuzumab ozogamicin 3 mg/m2 on days 4 and 8. Includes cohort 4 from the Phase 1 portion of the study.
Arm/Group | Phase 1 Dose-Finding Cohorts 1-3 | Phase 2/Selected Dose
Number analyzed (Participants) | 9 | 43
participants | 4 | 18

3. Secondary Outcome: Number of Participants With Complete Remission
Description: Efficacy Defined as Best Response Achieved During Study Treatment Measured by Complete Remission (CR) Rate
Time Frame: up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2/Selected Dose
Number analyzed (Participants) | 43
Participants | 18

4. Secondary Outcome: Disease Relapse
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2/Selected Dose
Number analyzed (Participants) | 18
Participants | 5

ADVERSE EVENTS:
Time Frame: Adverse events are collected from the start of treatment until 30 days after the last dose.
Groups:
- Phase 1 Dose-Finding: Patients receive vorinostat PO on days 1-9, azacitidine SC or IV over 10-40 minutes on days 1-7, and gemtuzumab ozogamicin IV over 2 hours on day 8. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Laboratory biomarker analysis: correlative studies
- Phase 2: Azacitidine 75 mg/m2 on days 1-7, vorinostat 400 mg qd on days 1-9, gemtuzumab ozogamicin 3 mg/m2 on days 4 and 8. Includes cohort 4 from the Phase 1 portion of the study.
  Laboratory biomarker analysis: correlative studies
Arm/Group | Phase 1 Dose-Finding | Phase 2
Serious Adverse Events (participants affected / at risk) | 6/15 | 13/43
Other Adverse Events (participants affected / at risk) | 9/15 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose-Finding (N=15) | Phase 2 (N=43)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
hypotension (Cardiac disorders) | 1 (1) | 2 (2)
infection with neutropenia (Infections and infestations) | 1 (2) | 1 (2)
febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
sepsis (Infections and infestations) | 0 (0) | 4 (4)
multi-organ failure (General disorders) | 0 (0) | 1 (1)
death, NOS (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose-Finding (N=15) | Phase 2 (N=43)
abdominal pain (General disorders) | 1 (1) | 5 (6)
acidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
blood chemistry changes (Metabolism and nutrition disorders) | 9 (67) | 43 (86)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 5 (5)
elevated liver function tests (Hepatobiliary disorders) | 6 (14) | 15 (32)
allergic reaction (Immune system disorders) | 0 (0) | 2 (3)
bleeding (Blood and lymphatic system disorders) | 4 (4) | 19 (19)
anemia (Blood and lymphatic system disorders) | 8 (11) | 25 (33)
anorexia (Metabolism and nutrition disorders) | 1 (1) | 23 (34)
anxiety (Psychiatric disorders) | 0 (0) | 7 (7)
aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 13 (17)
bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
cardiac chest pain (Cardiac disorders) | 0 (0) | 2 (2)
chills (General disorders) | 2 (2) | 19 (19)
colitis (Gastrointestinal disorders) | 0 (0) | 4 (4)
confusion (Psychiatric disorders) | 0 (0) | 8 (8)
constipation (Gastrointestinal disorders) | 5 (6) | 15 (18)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 16 (17)
depression (Psychiatric disorders) | 2 (3) | 4 (4)
infection (Infections and infestations) | 5 (9) | 37 (43)
diarrhea (Gastrointestinal disorders) | 5 (5) | 22 (26)
dizziness (Nervous system disorders) | 2 (3) | 11 (11)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 14 (14)
edema (General disorders) | 2 (2) | 11 (12)
prolonged QTc (Cardiac disorders) | 0 (0) | 4 (4)
erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
fatigue (General disorders) | 4 (5) | 29 (39)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 31 (44)
fever (General disorders) | 0 (0) | 16 (20)
pain (General disorders) | 3 (4) | 14 (15)
muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6)
headache (Nervous system disorders) | 2 (2) | 8 (9)
hypertension (Cardiac disorders) | 1 (1) | 9 (11)
hypotension (Cardiac disorders) | 2 (2) | 9 (9)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (9)
infusion reaction (Immune system disorders) | 0 (0) | 4 (5)
lymphopenia (Blood and lymphatic system disorders) | 4 (6) | 0 (0)
malaise (General disorders) | 0 (0) | 3 (3)
mucositis (Gastrointestinal disorders) | 0 (0) | 6 (7)
nausea (Gastrointestinal disorders) | 8 (10) | 33 (47)
neutropenia (Blood and lymphatic system disorders) | 3 (4) | 17 (26)
non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
thrombocytopenia (Blood and lymphatic system disorders) | 5 (6) | 25 (38)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
skin disorders (Skin and subcutaneous tissue disorders) | 3 (3) | 15 (15)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
sepsis (Infections and infestations) | 0 (0) | 9 (9)
vomiting (Gastrointestinal disorders) | 6 (8) | 17 (25)
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
leukopenia (Blood and lymphatic system disorders) | 6 (7) | 23 (32)
sinus tachycardia (Cardiac disorders) | 1 (1) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less